CLINICAL TRIAL: NCT02882399
Title: Shortystrap Effectiveness in the Treatment of the Pathology Pubic and Abdominal Pathology in Athletes
Acronym: Shortystrap
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-A01172-41; 35RC12_8971 (Other: CHU Rennes)
Record Dates: First submitted 2016-08-22; First posted 2016-08-29 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2016-08

CONDITIONS: Pubic and Abdominal Pathology
Keywords: athletes

ARMS (1):
- Shortystrap (Experimental)
  Interventions: Other: Shortystrap

INTERVENTIONS:
Other: Shortystrap

SUMMARY:
The pubic and abdominal pathology is common among athletes. It leads to a shutdown of physical activity for several months, and requires rehabilitative care, or surgery for a permanent cure. Shortystrap is designed to avoid surgery and allow the continuation of sports.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Sports practicing physical activity at least 3 hours per week
* Practicing a team sport with a major part of running (football, rugby, ...)
* Presenting a pubic and abdominal pathology for at least 4 weeks
* In primary consultation
* Age from 18 to 40 years
* Informed consent signed

Exclusion Criteria:

* Professional athlete
* Cyclist
* Having already received usual medical treatment (anti-inflammatory treatment and rest)
* Introducing another disease requiring treatment with NSAIDs
* Allergy neoprene
* Contraindications to performing MRI (claustrophobia, any metal device, pacemaker, etc.)
* Simultaneous participation in another biomedical research
* Major person under legal protection (backup justice, trusteeship, guardianship), person deprived of liberty.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-04-12 (Actual); Primary Completion 2015-08-20 (Actual); Study Completion 2015-11-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain using a scale Feretti | Day 15
  scale Feretti

SECONDARY OUTCOMES:
Evaluation of pain using a visual analog scale | Day 15, Day 30 and Day 60
  visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Pierrick GUILLEMOT, Md, Study Director — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France